CLINICAL TRIAL: NCT03248531
Title: A Phase 2 Multicenter, Investigator-Blind, Subject-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Pharmacokinetics of Bimekizumab in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Test the Efficacy, Safety and Pharmacokinetics of Bimekizumab in Subjects With Moderate to Severe Hidradenitis Suppurativa.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS0001; 2017-000892-10 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-14 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Bimekizumab; HS; Moderate to Severe HS
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bimekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bimekizumab (Experimental): Subjects will receive one Bimekizumab loading dose 1 and several Bimekizumab dose 2 applications.
  Interventions: Drug: Bimekizumab
- Adalimumab (Active Comparator): Subjects will receive one Adalimumab loading (dose 1) and several Adalimumab dose 2 and dose 3 applications.
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Subjects will receive several placebo applications to keep the blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab in different dosages (dose 1 and 2).
  Other Names: UCB4940
  Arms: Bimekizumab
Drug: Adalimumab — Adalimumab in different dosages (dose 1, 2 and 3).
  Other Names: Humira®
  Arms: Adalimumab
Other: Placebo — Placebo will be provided matching Bimekizumab.
  Arms: Placebo

SUMMARY:
Hidradenitis suppurativa (HS) is a painful, long-term skin condition that causes abscesses and scarring on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 to 70 years of age, inclusive) must have a diagnosis of HS for at least

  1 year prior to Baseline
* Stable HS for at least 2 months prior to Screening and also at the Baseline Visit
* Inadequate response to at least a 3-month study of an oral antibiotic for treatment of HS
* Total abscess and inflammatory nodule count >=3 at the Baseline Visit
* Subject must agree to daily use (and throughout the entirety of the study) of 1 pre-specified over-the-counter topical antiseptics on their HS lesions
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception up till 20 weeks after last administration of study drug and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to first dose
* Male subjects must be willing to use a method of contraception when sexually active, up till 20 weeks after the last administration of study medication

Exclusion Criteria:

* Prior treatment with anti-IL17s or participation in an anti-IL17 study
* Previously received anti-TNFs
* Subject requires, or is expected to require, opioid analgesics for any reason (excluding tramadol)
* Subject received prescription topical therapies for the treatment of HS within 14 days prior to the Baseline Visit
* Subject received systemic non-biologic therapies for HS with potential therapeutic impact for HS less than 28 days prior to Baseline Visit
* Draining fistula count >20 at the Baseline Visit
* Diagnosis of inflammatory conditions other than HS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1-844-599-2273 (UCB)
Locations (31):
- United States (11):
  - Hs0001 121, Los Angeles, California
  - Hs0001 119, Coral Gables, Florida
  - Hs0001 111, Orange, Florida
  - Hs0001 117, Tampa, Florida
  - Hs0001 112, Sandy Springs, Georgia
  - Hs0001 113, Boston, Massachusetts
  - Hs0001 115, Las Vegas, Nevada
  - Hs0001 126, Manhasset, New York
  - Hs0001 125, Chapel Hill, North Carolina
  - Hs0001 123, Hershey, Pennsylvania
  - Hs0001 120, Nashville, Tennessee
- Australia (5):
  - Hs0001 103, East Melbourne
  - Hs0001 101, Fremantle
  - Hs0001 104, Saint Leonards
  - Hs0001 100, Westmead
  - Hs0001 102, Woolloongabba
- Belgium (2):
  - Hs0001 203, Brussels
  - Hs0001 202, Liège
- Hs0001 300, Copenhagen, Denmark
- Germany (6):
  - Hs0001 408, Berlin
  - Hs0001 405, Bochum
  - Hs0001 407, Darmstadt
  - Hs0001 400, Dessau
  - Hs0001 404, Erlangen
  - Hs0001 406, Würzburg
- Hs0001 503, Athens, Greece
- Norway (2):
  - Hs0001 701, Harstad
  - Hs0001 700, Tromsø
- Russia (3):
  - Hs0001 901, Moscow
  - Hs0001 903, Saint Petersburg
  - Hs0001 900, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glatt S, Jemec GBE, Forman S, Sayed C, Schmieder G, Weisman J, Rolleri R, Seegobin S, Baeten D, Ionescu L, Zouboulis CC, Shaw S. Efficacy and Safety of Bimekizumab in Moderate to Severe Hidradenitis Suppurativa: A Phase 2, Double-blind, Placebo-Controlled Randomized Clinical Trial. JAMA Dermatol. 2021 Nov 1;157(11):1279-1288. doi: 10.1001/jamadermatol.2021.2905. PMID 34406364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2017 and concluded in February 2019.
Pre-assignment Details: The study included a Screening Period (≥ 2 weeks up to a maximum of 4 weeks prior to randomization), a Treatment Period (12 weeks), and a Safety Follow-Up (SFU) Visit (20 weeks after the last dose of investigational medicinal product (IMP)). Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received matching placebo subcutaneous (SC) injections at Baseline, followed by Week 2, 4, 5, 6, 7, 8, 9, and 10 to maintain study blinding.
- Adalimumab: Participants received one adalimumab 160 milligrams (mg) SC injection as loading dose started from Baseline, followed by adalimumab 80 mg SC injection at Week 2 and adalimumab 40 mg SC injections from Weeks 4 to 10. Participants also received matching placebo SC injection at Week 4, 6, 8 and 10 to maintain study blinding.
- Bimekizumab: Participants received one bimekizumab 640 mg SC injection as loading dose started from Baseline, followed by bimekizumab 320 mg SC injections at Weeks 2, 4, 6, 8 and 10. Participants also received matching placebo SC injections at Week 5, 7 and 9 to maintain study blinding.
Period: Overall Study
Arm/Group | Placebo | Adalimumab | Bimekizumab
Started (Completed screening period (2-4 Weeks) and Randomized) | 22 | 22 | 46
Completed Week 12 (Completed treatment period (12 Weeks)) | 19 | 18 | 42
Completed (Study completed (including safety follow-up period [20 weeks after last dose])) | 18 | 17 | 38
Not Completed | 4 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 5
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Sponsor Request | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all study participants randomized into the study.
Arm/Group | Placebo | Adalimumab | Bimekizumab | Total Title
Number analyzed (Participants) | 22 | 22 | 46 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 2
  Between 18 and 65 years | 21 | 22 | 44 | 87
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.5) | 31.0 (9.2) | 37.4 (11.9) | 36.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 30 | 63
  Male | 7 | 4 | 16 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 0 | 1
  Asian | 1 | 3 | 0 | 4
  Black or African American | 6 | 5 | 10 | 21
  White | 12 | 14 | 35 | 61
  Other or Mixed | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response as Measured by Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR was defined as at least a 50 % reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase from Baseline in abscess or draining fistula count. Results were based on a Bayesian logistic regression model where the number of responders were assumed to follow a binomial distribution. Participants with missing data at Week 12 were considered as nonresponders in the analysis. Posterior mean response rates and 95% credible intervals in each group are presented.
Time Frame: Week 12
Population: The Per-Protocol Set (PPS) was a subset of the Full Analysis Set (FAS), consisting of those study participants who had no important protocol deviations affecting the primary efficacy variable, as confirmed during a pre-analysis review prior to unblinding of the data (at each of the interim and final analyses).
Measure: Mean (95% Confidence Interval); unit: Percentage of responders
Groups:
- Placebo (PPS): Participants received matching placebo subcutaneous (SC) injections at Baseline, followed by Week 2, 4, 5, 6, 7, 8, 9, and 10 to maintain study blinding, forming the Per-Protocol Set (PPS).
- Adalimumab (PPS): Participants received one adalimumab 160 milligrams (mg) SC injection as loading dose started from Baseline, followed by adalimumab 80 mg SC injection at Week 2 and adalimumab 40 mg SC injections from Weeks 4 to 10. Participants also received matching placebo SC injection at Week 4, 6, 8 and 10 to maintain study blinding, forming the PPS.
- Bimekizumab (PPS): Participants received one bimekizumab 640 mg SC injection as loading dose started from Baseline, followed by bimekizumab 320 mg SC injections at Weeks 2, 4, 6, 8 and 10. Participants also received matching placebo SC injections at Week 5, 7 and 9 to maintain study blinding, forming the PPS.
Arm/Group | Placebo (PPS) | Adalimumab (PPS) | Bimekizumab (PPS)
Number analyzed (Participants) | 20 | 20 | 44
Percentage of responders | 26.1 [13.8 to 40.5] | 59.5 [44.2 to 73.9] | 57.3 [42.4 to 71.4]
Statistical Analysis 1: Comparison: Placebo (PPS) vs Bimekizumab (PPS); Results were based on a Bayesian logistic regression model where the number of responders were assumed to follow a binomial distribution. Treatment and Baseline Hurley Stage were included as predictors in the model. 95% credible intervals were presented for the bimekizumab (BKZ) vs placebo (PBO) comparison; Test type: Other; Regression, Logistic; Mean posterior difference = 31.2, 95% CI 2-sided [11.0 to 50.4], Standard Deviation 10.1
Statistical Analysis 2: Comparison: Adalimumab (PPS) vs Bimekizumab (PPS); Results were based on a Bayesian logistic regression model where the number of responders were assumed to follow a binomial distribution. Treatment and Baseline Hurley Stage were included as predictors in the model. 60% credible intervals were presented for the BKZ vs adalimumab (ADA) comparison; Test type: Other; Regression, Logistic; Mean posterior difference = -2.2, 60% CI 2-sided [-11.2 to 6.6], Standard Deviation 10.6
Statistical Analysis 3: Comparison: Placebo (PPS) vs Bimekizumab (PPS); Results were based on a Bayesian logistic regression model where the number of responders were assumed to follow a binomial distribution. Treatment and Baseline Hurley Stage were included as predictors in the model; Test type: Other; Regression, Logistic; Pr [Diff>0%] (%) = 99.8
Statistical Analysis 4: Comparison: Adalimumab (PPS) vs Bimekizumab (PPS); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Logistic; Pr[Diff > 0%](%) = 42.1

2. Secondary Outcome: Bimekizumab Plasma Concentration at Day 1 (Prior to First Dose)
Description: Plasma concentration of Bimekizumab was expressed in nanograms per milliliter (ng/mL). Values Below Limit of Quantification (BLQ) were replaced by value of Lower Limit of Quantification (LLOQ) divided by 2 (75 ng/mL) in calculations of Means and Coefficient of Variations (CVs).
Time Frame: Day 1 (Prior to first dose)
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had at least 1 quantifiable postdose plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Bimekizumab (PK-PPS): Participants received one bimekizumab 640 mg SC injection as loading dose started from Baseline, followed by bimekizumab 320 mg SC injections at Weeks 2, 4, 6, 8 and 10. Participants also received matching placebo SC injections at Week 5, 7 and 9 to maintain study blinding, forming the Pharmacokinetic Per-Protocol Set (PK-PPS).
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 46
ng/mL | NA (NA) — Here, NA signifies that geometric means and geometric CVs were only calculated if at least 2/3 of the concentrations were above lower limit of quantification (LLOQ).

3. Secondary Outcome: Bimekizumab Plasma Concentration at Week 2
Description: Plasma concentration of Bimekizumab was expressed in ng/mL. Values BLQ were replaced by value of LLOQ/2 (75 ng/mL) in calculations of Means and CVs.
Time Frame: Week 2
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had at least 1 quantifiable postdose plasma concentration. Here, number of participants analyzed included all participants who were evaluable for this Outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Bimekizumab (PK-PPS): Participants received one bimekizumab 640 mg SC injection as loading dose started from Baseline, followed by bimekizumab 320 mg SC injections at Weeks 2, 4, 6, 8 and 10. Participants also received matching placebo SC injections at Week 5, 7 and 9 to maintain study blinding, forming the PK-PPS.
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 45
ng/mL | 24086.4 (56.4)

4. Secondary Outcome: Bimekizumab Plasma Concentration at Week 4
Description: as for outcome 3
Time Frame: Week 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 46
ng/mL | 26572.6 (57.6)

5. Secondary Outcome: Bimekizumab Plasma Concentration at Week 8
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 43
ng/mL | 30222.6 (54.5)

6. Secondary Outcome: Bimekizumab Plasma Concentration at Week 12
Description: as for outcome 3
Time Frame: Week 12
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 42
ng/mL | 25319.0 (116.8)

7. Secondary Outcome: Bimekizumab Plasma Concentration at Week 30
Description: as for outcome 3
Time Frame: Week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 35
ng/mL | NA (NA) — Here, NA signifies that geometric means and geometric CVs were only calculated if at least 2/3 of the concentrations were above lower limit of quantification (LLOQ).

8. Secondary Outcome: Percentage of Participants With at Least One Adverse Event During the Study
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Screening to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Participants received matching placebo subcutaneous (SC) injections at Baseline, followed by Week 2, 4, 5, 6, 7, 8, 9, and 10 to maintain study blinding, forming the Safety Set (SS).
- Adalimumab (SS): Participants received one adalimumab 160 milligrams (mg) SC injection as loading dose started from Baseline, followed by adalimumab 80 mg SC injection at Week 2 and adalimumab 40 mg SC injections from Weeks 4 to 10. Participants also received matching placebo SC injection at Week 4, 6, 8 and 10 to maintain study blinding, forming the SS.
- Bimekizumab (SS): Participants received one bimekizumab 640 mg SC injection as loading dose started from Baseline, followed by bimekizumab 320 mg SC injections at Weeks 2, 4, 6, 8 and 10. Participants also received matching placebo SC injections at Week 5, 7 and 9 to maintain study blinding, forming the SS.
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 21 | 21 | 46
percentage of participants | 61.9 | 71.4 | 71.7

9. Secondary Outcome: Percentage of Participants With at Least One Adverse Event Categorized by Maximum Severity During the Study
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. To record the intensity of an AE Investigator used the following criteria: Mild: the study participant was aware of sign or symptom (syndrome), but it did not interfere with his/her usual activities and/or was of no clinical consequence; Moderate: AE interfered with the usual activities of the study participant or it was of some clinical consequence; Severe: the study participant was unable to work normally or to carry out his/her usual activities, or the AE was of definite clinical consequence.
Time Frame: From Screening to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 21 | 21 | 46
percentage of participants
  Mild | 47.6 | 66.7 | 63.0
  Moderate | 33.3 | 42.9 | 39.1
  Severe | 4.8 | 9.5 | 6.5

10. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event During the Study
Description: A serious adverse event (SAE) was any untoward medical occurrence that at any dose: Resulted in death, was life-threatening, required in patient hospitalization or prolongation of existing hospitalisation, was a congenital anomaly or birth defect, was an infection that required treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may have jeopardised the patients, or may have required medical or surgical intervention to prevent any of the above.
Time Frame: From Screening to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 21 | 21 | 46
percentage of participants | 9.5 | 4.8 | 4.3

11. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event Categorized by Severity During the Study
Description: A serious adverse event (SAE) was any untoward medical occurrence that at any dose: Resulted in death, was life-threatening, required in patient hospitalization or prolongation of existing hospitalization, was a congenital anomaly or birth defect, was an infection that required treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may have jeopardised the patients, or may have required medical or surgical intervention to prevent any of the above. To record the intensity of an AE Investigator used the following criteria: Mild: study participant was aware of sign or symptom (syndrome), but it did not interfere with his/her usual activities and/or was of no clinical consequence; Moderate: AE interfered with usual activities of study participant or it was of some clinical consequence; Severe: the study participant was unable to work normally or to carry out his/her usual activities, or the AE was of definite clinical consequence.
Time Frame: From Screening to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 21 | 21 | 46
percentage of participants
  Mild | 0 | 4.8 | 0
  Moderate | 4.8 | 0 | 0
  Severe | 4.8 | 4.8 | 4.3

12. Secondary Outcome: Percentage of Participants That Withdrew Due to Adverse Events During the Study
Description: as for outcome 8
Time Frame: From Screening to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 21 | 21 | 46
percentage of participants | 0 | 0 | 2.2

13. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Vital Signs (Blood Pressure)
Description: Blood pressure was measured in millimeters of mercury (mmHg).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP. Here, number of participants analyzed included all participants who were evaluable for this Outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 19 | 38
mmHg
  Systolic Blood Pressure | -2.9 (14.8) | 4.5 (14.5) | -0.4 (13.8)
  Diastolic Blood Pressure | -1.8 (8.4) | -0.6 (9.1) | -2.2 (11.2)

14. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Vital Signs (Pulse Rate)
Description: Pulse rate was measured in beats per minute (beats/min).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 19 | 38
beats/min | -1.4 (10.2) | -1.8 (10.8) | -1.6 (10.8)

15. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Body Weight
Description: Body weight was measured in kilograms (kg).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 19 | 38
kg | 0.90 (7.39) | 1.82 (3.94) | 0.42 (6.89)

16. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in ECG Parameters (ECG Mean Heart Rate)
Description: Electrocardiogram (ECG) Mean Heart Rate was measured in beats/min.
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 15 | 37
beats/min | -2.1 (12.4) | -2.1 (11.1) | 1.5 (10.1)

17. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in ECG Parameters (PR Interval, QRS Duration, QT Interval, QTcF Interval)
Description: PR Interval, QRS duration, QT interval and QT corrected for heart rate using Fridericia's correction (QTcF) Interval were measured in milliseconds (msec).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 15 | 37
msec
  PR Interval | 0.8 (18.8) | 2.4 (10.5) | 3.6 (18.7)
  QRS duration | -0.3 (7.1) | 0.2 (5.2) | 0.6 (7.4)
  QT interval | 4.8 (20.2) | 4.2 (26.7) | 1.8 (27.7)
  QTcF Interval | -11.7 (49.9) | -0.3 (14.4) | 2.4 (12.7)

18. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes)
Description: Erythrocytes was measured in number of red blood cells per liter (10^12/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^12 red blood cells per liter
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
10^12 red blood cells per liter | 0.144 (0.349) | -0.151 (0.416) | -0.013 (0.274)

19. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Hematocrit)
Description: Hematocrit was measured in volume percentage (%) of red blood cells in blood.
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: volume % of red blood cells
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
volume % of red blood cells | 2.01 (2.83) | -0.81 (4.30) | 0.39 (2.69)

20. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Hemoglobin, Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration)
Description: Hemoglobin, erythrocytes mean corpuscular hemoglobin (HGB) concentration were measured in grams per liter (g/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
g/L
  Hemoglobin | 5.3 (11.6) | -3.7 (11.6) | 1.1 (7.6)
  Erythrocytes mean corpuscular HGB | -1.4 (16.2) | -2.6 (13.4) | -0.2 (13.2)

21. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes Mean Corpuscular Hemoglobin (HGB))
Description: Erythrocytes mean corpuscular hemoglobin (HGB) was measured in picograms (pg).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
picograms (pg) | 0.29 (0.76) | 0.21 (0.78) | 0.30 (0.99)

22. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes Mean Corpuscular Volume)
Description: Erythrocytes mean corpuscular volume was measured in femtoliters (fL).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
femtoliters (fL) | 1.49 (2.95) | 1.36 (3.21) | 1.04 (4.03)

23. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Platelets)
Description: Platelets was measured in number of platelets per liter (10^9/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
10^9 platelets per liter | -17.4 (38.7) | 2.3 (61.6) | -19.2 (51.4)

24. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Leukocytes, Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils)
Description: Leukocytes, basophils, eosinophils, lymphocytes, monocytes and neutrophils were measured in number of white blood cells per liter (10^9/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: 10^9 white blood cells per liter
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
10^9 white blood cells per liter
  Leukocytes | -0.281 (2.621) | -0.114 (2.997) | -0.122 (2.308)
  Basophils | 0.009 (0.026) | 0.033 (0.077) | 0.015 (0.048)
  Eosinophils | 0.007 (0.077) | -0.012 (0.100) | 0.002 (0.056)
  Lymphocytes | 0.029 (0.812) | 0.241 (0.682) | 0.038 (0.570)
  Monocytes | 0.072 (0.420) | -0.032 (0.322) | 0.060 (0.192)
  Neutrophils | -0.396 (2.076) | -0.341 (2.460) | -0.240 (2.234)

25. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes)
Description: Basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes and neutrophils/leukocytes were measured in percentages (%).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: % of white blood cells per leukocytes
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 18 | 33
% of white blood cells per leukocytes
  Basophils/leukocytes | 0.13 (0.23) | 0.42 (0.93) | 0.13 (0.65)
  Eosinophils/leukocytes | -0.12 (1.92) | -0.03 (1.09) | 0.12 (1.12)
  Lymphocytes/leukocytes | 1.43 (5.47) | 2.04 (6.73) | 2.04 (8.07)
  Monocytes/leukocytes | 0.49 (4.35) | -0.20 (2.79) | 1.00 (2.17)
  Neutrophils/leukocytes | -1.93 (6.84) | -2.24 (7.50) | -3.29 (9.55)

26. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Bicarbonate, Chloride, Potassium, Sodium, Calcium, Magnesium, Urea Nitrogen, Cholesterol, Glucose)
Description: Bicarbonate, chloride, potassium, sodium, calcium, magnesium, urea nitrogen, cholesterol and glucose were measured in millimoles per liter (mmol/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 15 | 19 | 36
mmol/L
  Bicarbonate | -0.1 (2.1) | 0.7 (2.8) | 0.6 (2.3)
  Chloride | 0.9 (1.5) | 1.3 (2.4) | 0.1 (2.2)
  Potassium | -0.13 (0.79) | -0.09 (0.37) | 0.03 (0.41)
  Sodium | 0.4 (1.5) | 0.4 (1.6) | 0.1 (2.2)
  Calcium | 0.027 (0.065) | 0.008 (0.144) | 0.067 (0.095)
  Magnesium | -0.029 (0.087) | -0.027 (0.052) | -0.009 (0.081)
  Urea nitrogen | 0.00 (1.46) | -0.43 (1.37) | 0.29 (1.79)
  Cholesterol | -0.311 (0.667) | -0.177 (0.634) | 0.157 (0.585)
  Glucose | 1.049 (1.835) | 0.436 (2.990) | 0.439 (2.212)

27. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Creatinine, Bilirubin, Urate)
Description: Creatinine, bilirubin, and urate were measured in micromols per liter (μmol/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP. Here, number of participants analyzed included all participants who were evaluable for this Outcome measure and 'n' (Number analyzed) signifies participants who were evaluable for each parameter.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 15 | 19 | 36
μmol/L
  Creatinine | -1.73 (9.92) | -1.72 (9.04) | 3.84 (9.22)
  Bilirubin: number analyzed (Participants) | 15 | 19 | 34
  Bilirubin | 0.17 (3.48) | -1.38 (3.04) | 0.18 (4.35)
  Urate: number analyzed (Participants) | 15 | 19 | 34
  Urate | 8.7 (52.2) | -8.9 (50.5) | 1.5 (43.1)

28. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (C Reactive Protein High Sensitivity)
Description: C reactive protein high sensitivity was measured in milligrams per liter (mg/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 15 | 19 | 36
mg/L | -2.801 (16.851) | -4.865 (21.863) | -2.810 (10.853)

29. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, Lactate Dehydrogenase)
Description: Alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase, lactate dehydrogenase were measured in units per liter (U/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 15 | 19 | 36
U/L
  Alanine aminotransferase: number analyzed (Participants) | 15 | 19 | 34
  Alanine aminotransferase | -3.3 (8.3) | -3.6 (9.8) | 3.6 (23.8)
  Alkaline phosphatase | -2.0 (12.2) | -2.4 (13.5) | -3.4 (11.6)
  Aspartate aminotransferase | -0.6 (3.6) | -1.0 (5.8) | 2.0 (13.3)
  Gamma glutamyl transferase | -2.0 (9.5) | 1.8 (14.2) | 2.3 (10.1)
  Lactate dehydrogenase | -17.0 (29.9) | -16.3 (35.6) | -12.8 (61.8)

30. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine pH)
Description: Urine pH was measured on a pH scale.
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 16 | 31
pH | -0.43 (0.98) | -0.25 (0.55) | -0.03 (0.69)

31. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine Albumin)
Description: Urine albumin was measured in milligrams per liter (mg/L).
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 15 | 18 | 34
mg/L | 50.80 (211.30) | -28.25 (121.29) | 0.49 (19.92)

32. Secondary Outcome: Number of Participants Who Shifted From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine Glucose)
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP. Here, number of participants analyzed included all the participants with non-missing urinalysis results at Baseline and at Week 30 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 16 | 31
Participants
  Baseline Low - Week 30 Low | 0 | 0 | 0
  Baseline Low - Week 30 Normal | 0 | 0 | 0
  Baseline Low - Week 30 High | 0 | 0 | 0
  Baseline Normal - Week 30 Low | 0 | 0 | 0
  Baseline Normal - Week 30 Normal | 12 | 14 | 28
  Baseline Normal - Week 30 High | 1 | 1 | 0
  Baseline High - Week 30 Low | 0 | 0 | 0
  Baseline High - Week 30 Normal | 0 | 1 | 1
  Baseline High - Week 30 High | 1 | 0 | 2

33. Secondary Outcome: Number of Participants Who Shifted From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine Leukocyte Esterase)
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 14 | 16 | 31
Participants
  Baseline Low - Week 30 Low | 0 | 0 | 0
  Baseline Low - Week 30 Normal | 0 | 0 | 0
  Baseline Low - Week 30 High | 0 | 0 | 0
  Baseline Normal - Week 30 Low | 0 | 0 | 0
  Baseline Normal - Week 30 Normal | 8 | 9 | 19
  Baseline Normal - Week 30 High | 2 | 0 | 6
  Baseline High - Week 30 Low | 0 | 0 | 0
  Baseline High - Week 30 Normal | 2 | 3 | 6
  Baseline High - Week 30 High | 2 | 4 | 0

34. Secondary Outcome: Number of Participants Who Shifted From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine Bacteria)
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 3 | 6 | 2
Participants
  Baseline Low - Week 30 Low | 0 | 0 | 0
  Baseline Low - Week 30 Normal | 0 | 0 | 0
  Baseline Low - Week 30 High | 0 | 0 | 0
  Baseline Normal - Week 30 Low | 0 | 0 | 0
  Baseline Normal - Week 30 Normal | 0 | 0 | 0
  Baseline Normal - Week 30 High | 0 | 0 | 0
  Baseline High - Week 30 Low | 0 | 0 | 0
  Baseline High - Week 30 Normal | 0 | 0 | 0
  Baseline High - Week 30 High | 3 | 6 | 2

35. Secondary Outcome: Number of Participants Who Shifted From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (Urine Erythrocytes)
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 3 | 1 | 1
Participants
  Baseline Low - Week 30 Low | 0 | 0 | 0
  Baseline Low - Week 30 Normal | 0 | 0 | 0
  Baseline Low - Week 30 High | 0 | 0 | 0
  Baseline Normal - Week 30 Low | 0 | 0 | 0
  Baseline Normal - Week 30 Normal | 1 | 0 | 1
  Baseline Normal - Week 30 High | 0 | 0 | 0
  Baseline High - Week 30 Low | 0 | 0 | 0
  Baseline High - Week 30 Normal | 0 | 0 | 0
  Baseline High - Week 30 High | 2 | 1 | 0

36. Secondary Outcome: Number of Participants Who Shifted From Baseline Until Safety Follow-up Visit in Physical Examination
Time Frame: From Baseline to Safety Follow-Up (Week 30)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose (full or partial) of IMP. Here, number of participants analyzed included all the participants with a normal/at least one abnormal physical examination assessment and with non-missing physical examination assessment results at Baseline and at Week 30 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 18 | 19 | 38
Participants
  Baseline Normal - Week 30 Normal | 14 | 15 | 28
  Baseline Normal - Week 30 Abnormal | 1 | 2 | 5
  Baseline Abnormal - Week 30 Normal | 1 | 1 | 1
  Baseline Abnormal - Week 30 Abnormal | 2 | 1 | 4

37. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Day 1
Description: The overall status of a study participant was 'Positive' if at any post-Baseline visit the result was positive. Percentages were based on the number of study participants with a non-missing measurement, from samples that did not contain BKZ concentration levels above the drug tolerance, at the visit.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 46
percentage of participants | 4.3

38. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Week 2
Description: as for outcome 37
Time Frame: Week 2
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had at least 1 quantifiable postdose plasma concentration. Here, the number of participants analyzed included all participants who were evaluable with a non-missing measurement for this Outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 45
percentage of participants | 4.4

39. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Week 4
Description: as for outcome 37
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 46
percentage of participants | 4.3

40. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Week 8
Description: as for outcome 37
Time Frame: Week 8
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 42
percentage of participants | 0

41. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Week 12
Description: as for outcome 37
Time Frame: Week 12
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 42
percentage of participants | 9.5

42. Secondary Outcome: Percentage of Participants With Positive Bimekizumab Anti-drug Antibody (ADA) Concentration at Week 30
Description: as for outcome 37
Time Frame: Week 30
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab (PK-PPS)
Number analyzed (Participants) | 36
percentage of participants | 13.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Baseline (Day 1) until the Safety Follow-Up Visit (Week 30)
Description: A treatment-emergent AE (TEAE) was defined as any AE with a start date/time at the time of or after the first dose of IMP up until 140 days after the last dose of IMP.
Arm/Group | Placebo (SS) | Adalimumab (SS) | Bimekizumab (SS)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/21 | 2/46
Other Adverse Events (participants affected / at risk) | 5/21 | 12/21 | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=21) | Adalimumab (SS) (N=21) | Bimekizumab (SS) (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=21) | Adalimumab (SS) (N=21) | Bimekizumab (SS) (N=46)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (4)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (3)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 3 (4)
Hidradenitis (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 8 (9)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT03248531/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT03248531/SAP_001.pdf